CLINICAL TRIAL: NCT00366262
Title: A Randomized, Double-Blind, Parallel Group Study To Compare The 7-Day Gastrointestinal Safety of 2 Doses of PLA-695 To That Of Placebo And Naproxen
Brief Title: Study Evaluating the Gastrointestinal Safety of PLA-695 Compared to Placebo and Naproxen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3175A1-103
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Health
MeSH Terms: interventions — PLA-695; Naproxen

INTERVENTIONS:
Drug: PLA-695
Drug: Naproxen
Drug: Placebo

SUMMARY:
The purpose of this study is to provide an initial assessment of the gastrointestinal safety of a 7-day regimen of PLA-695 compared to placebo or naproxen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women of nonchildbearing potential, aged 18 to 60 years.

Exclusion Criteria:

* Abnormal baseline endoscopy.
* Positive Helicobacter pylori serology.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-06; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The rate of erosions and ulcers present after 7 days of treatment for PLA-65 will be compared to placebo and naproxen.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Houston, Texas, United States